CLINICAL TRIAL: NCT05398653
Title: A Multicenter, Randomized, Controlled, Open Phase Ib/ Ⅱ Study Evaluating the Efficacy and Safety of Recombinant Humanized Monoclonal Antibody MIL62 Injection in the Treatment of Primary Membranous Nephropathy.
Brief Title: A Phase Ib/ Ⅱ Clinical Study of MIL62 in Primary Membranous Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIL62-CT206
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIL62(600mg) (Experimental)
  Interventions: Drug: MIL62
- Ciclosporin (Active Comparator)
  Interventions: Drug: Cyclosporine
- MIL62(1000mg) (Experimental)
  Interventions: Drug: MIL62

INTERVENTIONS:
Drug: MIL62 — A 600 mg intravenous (IV) infusion of MIL62 will be administered on Week 1 Day 1 and Week 3 Day 1. If treatment response is observed, additional doses will be administered on Week 25 Day 1 and Week 27 Day 1. According to the protocol amendment in June 2023, some patients also received MIL62 treatment on Week 53 Day 1.
  Arms: MIL62(600mg)
Drug: Cyclosporine — Participants will receive Cyclosporine at a starting oral dose 3.5 mg/kg/d, divided into 2 doses, try to give every 12 hours. The dose was adjusted according to the blood concentration of cyclosporine monitored every 2 weeks ±3 days until the target blood concentration of 125~175 ng/ mL was reached. Optimized cyclosporine dose will be maintained for a maximum 52 weeks dependent on response and then tapered over 8 weeks.
  Arms: Ciclosporin
Drug: MIL62 — A 1000 mg intravenous (IV) infusion of MIL62 will be administered on Week 1 Day 1 and Week 3 Day 1. If treatment response is observed, additional doses will be administered on Week 25 Day 1 and Week 27 Day 1. According to the protocol amendment in June 2023, some patients also received MIL62 treatment on Week 53 Day 1.
  Arms: MIL62(1000mg)

SUMMARY:
This study was divided into two stages. In the first stage (Phase Ib), 30 subjects were randomly divided into MIL62 600mg, MIL62 1000mg and cyclosporine groups at a ratio of 1:1:1, with 10 subjects in each group. Tolerance to MIL62 was evaluated within 4 weeks after the first administration. If the overall safety is determined by the investigator and sponsor to be tolerable to MIL62, phase II enrollment will be initiated.

The second stage(Phase II) was also randomly divided into MIL62 600mg, MIL62 1000mg and cyclosporine groups according to the ratio of 1:1:1, 20 subjects in each group, to evaluate the efficacy of MIL62 and cyclosporine in the treatment of primary membranous nephropathy. Eligible subjects in both phases received treatment and follow-up for a total of 104 weeks. The primary efficacy endpoints were the 12-week immune remission rate and the 24-week overall remission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, ≥18 years of age;
2. Diagnosis of primary membranous nephropathy (pMN) according to renal biopsy prior to or during screening；
3. Screening 24-hour urinary protein >= 5 g after best supportive care for >= 3 months prior to screening or screening 24-hour urinary protein > 3.5 g after best supportive care for >= 6 months prior to screening, or Screening 24-hour urinary protein > 3.5 g with at least one high-risk factor defined by the protocol;
4. Estimated glomerular filtration rate (eGFR ) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula ≥40 mL/min/1.73 m^2；
5. Sufficient organ function;
6. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Participants with a secondary cause of MN
2. Cyclosporine resistance
3. Urine protein decreased by > 50% within 6 months before screening
4. Received treatment drugs for membranous nephropathy
5. Concomitant with other serious diseases
6. Received live vaccination, major surgery (excluding diagnostic procedures), and participated in other clinical trials within 28 days prior to receiving the first study drug
7. Patients who are positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb), with HBV DNA levels above the normal range (HBsAg and/or HBcAb-positive patients require regular HBV DNA testing); patients positive for hepatitis C virus (HCV) antibodies; or patients with a positive human immunodeficiency virus (HIV) serology
8. Participants with CD4+ T lymphocyte count < 300 cells/μL
9. Those who have a clear history of tuberculosis or have received anti- tuberculosis treatment
10. Participants with known history of severe allergic reactions to humanized monoclonal antibodies, MIL62, or Cyclosporine
11. Breastfeeding or pregnant women
12. Childbearing potential and unwillingness or impossibility to comply with a scientifically acceptable birth-control method
13. Other conditions unsuitable for participation in this study determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Stage 1: The Tolerability and Safety of MIL62 in Participants with Primary Membranous Nephropathy | up to 2 year after enrollment
  Evaluation of the Tolerability and Safety of MIL62 in Participants with pMN.The tolerance is defined as the occurrence of CTCAE 5.0 Grade ≥3 adverse events within 28 days after the first dose of MIL62.Safety assessments included adverse events, vital signs, physical examinations, laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status and 12-lead electrocardiograms (ECG) during the study period.
Stage 1 and Stage 2: The 12-week immune remission rate in the anti-PLA2R antibody-positive population. | Week 12
  The proportion of participants who achieved immune remission(Anti-PLA2R antibody<14RU/mL) at week 12.
Stage 1 and Stage 2:The 24-week overall remission rate (ORR) | week 24
  The proportion of participants who achieved overall remission (complete and partial remission) at week 24.

SECONDARY OUTCOMES:
Stage 2: The immune remission rate at week 24, 52, 76, and 104. | Week 24, 52, 76 and 104
  The proportion of participants who achieved immune remissionat week 24, 52, 76, 104.
Stage 2: The complete remission rate (CRR) and partial remission rate (PRR) at week 24. | Week 24
  The proportion of participants who achieved complete remission (CR) and partial remission (PR) at week 24.
Stage 2:The CRR, PRR and ORR at week 52, 76, 104. | Week 52, 76, 104
  The proportion of participants who achieved CR、PR and overall remission (OR) at week 52,76,104.
Stage 2: Time to CR and OR | up to 104 weeks
Stage 2:The duration of CR and OR | up to 104 weeks
Stage 2: Change in anti-PLA2R antibody | up to 104 weeks
Stage 2: Change in eGFR | up to 104 weeks
Stage 2: Change in 24-hour urine protein | up to 104 weeks
Stage 2: Percentage of Participants with Adverse Events (AEs) | up to 104 weeks
  Severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Stage 2: Percentage of participants with AEs of Special Interest (AESIs) | up to 104 weeks
Stage 2: Peripheral B-cell Counts at Specified Timepoints. | up to 104 weeks
Stage 2: Incidence of ADAs during the study | up to 104 weeks
Stage 2: Pharmacokinetic(PK) Parameters during the study: Area Under the Curve(AUC) | up to 104 weeks
Stage 2: Pharmacokinetic(PK) Parameters during the study:Maximum Concentration(Cmax) | up to 104 weeks
Stage 2: Pharmacokinetic(PK) Parameters during the study: t1/2 | up to 104 weeks
Stage 2: Pharmacokinetic(PK) Parameters during the study: Volume of Distribution (Vd) | up to 104 weeks
Stage 2: Pharmacokinetic(PK) Parameters during the study: Clearance(CL) | up to 104 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China